CLINICAL TRIAL: NCT05229809
Title: Yiqi Wenyang Jiedu Prescription in the Prevention and Treatment of Postoperative Metastasis and Recurrence of Gastric Cancer：A Randomized, Double-blind, Controlled and Multi-center Clinical Study
Brief Title: Clinical Trial of Yiqi Wenyang Jiedu Prescription in the Prevention and Treatment of Postoperative Metastasis and Recurrence of Gastric Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jie Li (Other)
Responsible Party: Sponsor-Investigator, Jie Li, Assistant Dean, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI2021A01802
Record Dates: First submitted 2022-01-15; First posted 2022-02-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Gastric Carcinoma
Keywords: Postoperative gastric cancer; Yiqi Wenyang Jiedu prescription; Chinese Herbal Medicine; Randomized Controlled Trial; 2-year disease-free survival rate
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yiqi Wenyang Jiedu prescription Group (Experimental)
  Interventions: Drug: Yiqi Wenyang Jiedu prescription
- Simulation agent of Yiqi Wenyang Jiedu prescription Group (Placebo Comparator)
  Interventions: Drug: Simulation agent of Yiqi Wenyang Jiedu prescription

INTERVENTIONS:
Drug: Yiqi Wenyang Jiedu prescription — The dosage form of the test drug is granule. Patients need to take 2 small packets in the morning and 2 small packets in the evening. The medicine needs to be melted in hot water before being taken. Every 4 weeks is a course of treatment, a total of 6 courses,The patients were followed up to 3 years after gastric cancer surgery.
  Arms: Yiqi Wenyang Jiedu prescription Group
Drug: Simulation agent of Yiqi Wenyang Jiedu prescription — It is prepared from maltodextrin and food coloring. The raw materials of maltodextrin conform to the relevant provisions of excipients - maltodextrin in the fourth part of Chinese Pharmacopoeia 2015 edition. Food coloring includes caramel coloring, egg yolk coloring and milk chocolate brown pigment, all of which are edible grade ingredients. Patients need to take 2 small packets in the morning and 2 small packets in the evening. The medicine needs to be melted in hot water before being taken. Every 4 weeks is a course of treatment, a total of 6 courses,The patients were followed up to 3 years after gastric cancer surgery.
  Arms: Simulation agent of Yiqi Wenyang Jiedu prescription Group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Yiqi Wenyang Jiedu prescription for postoperative gastric cancer.

DETAILED DESCRIPTION:
This study include a multicenter, randomized, double-blind, placebo, parallel controlled clinical trial.The randomized clinical trial will enroll approximately 212 patients. Participants will be randomly divided into experimental (n=106) and control groups (n=106).Patients in the experimental group was treated with Yiqiuyang Jiedu prescription within 6-8 months after radical gastroctomy and after the completion of standard regimen (XELOX and SOX) for at least 6 cycles of adjuvant chemotherapy. Patients in the control group will receive the placebo.The primary endpoint is 2-year DFS (Disease-free survival) rate after surgery, that refers to the proportion of patients who do not have recurrence, metastasis or death (from any cause) within 2 years after surgery. The research protocol was approved by the relevant ethics committees, and the study was conducted according to the Declaration of Helsinki and Good Clinical Practice guidelines. Patients gave written informed consent to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. The non-esophagogastric junction gastric cancer of stage II-III that met the diagnostic criteria, and no tumor recurrence and metastasis was determined by imaging;
2. Within 6-8 months after radical gastrectomy for gastric cancer (R0), adjuvant chemotherapy of standard regimen (XELOX and SOX) has been completed for at least 6 cycles;
3. ECOG score 0-2;
4. 18-75 years old, male or female;
5. The expected survival time is ≥3 months;
6. Voluntary participation in the study, signing informed consent, good compliance with follow-up.

Exclusion Criteria:

1. Patients with other primary tumors;
2. Gastric cancer patients were pathologically diagnosed as adenosquamous carcinoma, with lymphoid stromal carcinoma (medullary carcinoma), hepatoid adenocarcinoma, squamous cell carcinoma, signed-ring cell carcinoma, undifferentiated carcinoma, gastric neuroendocrine tumor, gastric mesenchymal tumor, gastric malignant lymphoma and other gastric malignancies;
3. Patients who had previously received preoperative neoadjuvant chemotherapy;
4. Patients with past or current targeted drug therapy;
5. Patients undergoing previous or ongoing gastric radiotherapy;
6. Patients with past or ongoing tumor immunotherapy;
7. Mental patients;
8. Patients with serious and uncontrolled organic diseases or infections, such as decompensated heart, lung and renal failure, which lead to intolerance of chemotherapy;
9. Patients who received clinical trials of small molecule drugs within 28 days or large molecule drugs within 3 months;
10. Patients who are known to be allergic or intolerant to the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival rate | The day of surgery until the second year.
  Refers to the proportion of patients who did not experience recurrence, metastasis or death (from any cause) within 2 years after surgery.

SECONDARY OUTCOMES:
Disease-free survival | Randomization until disease recurrence, metastasis, death (from any cause) , or 36 months after surgery, whichever occurs first.
  It is the time from randomization to tumor progression or death (from any cause).
Overall survival | Randomization until death (from any cause) or 36 months after surgery, whichever occurs first.
  It is the time from randomization to death (from any cause).
Cumulative annual recurrence and metastasis rate for 1-3 years | The day of surgery until the once, second and third year.
  Refers to the proportion of patients with recurrence and metastasis within 1-3 years from the day of surgery.
Cumulative annual survival rate for 1-3 years | The day of surgery until the once, second and third year.
  Refers to the proportion of patients with survical within 1-3 years from the day of surgery.
Indexes related to fat distribution | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  Total Fat Area, Visceral Fat Area and Subcutaneous Fat Area. They measure fat area on cross-sectional images using plain CT scanning.
Visceral Adiposity Index | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  It is a new assessment of visceral fat based on waist circumference (WC), BMI, triglyceride (TG) and HDL.
  Male VAI = during [WC/(39.68 + 1.88 x BMI)] * (TG / 1.03) * (1.31 / HDL). Female VAI = during [WC/(36.58 + 1.89 x BMI)] * (TG / 0.81) * (1.52 / HDL).
Tumor marker | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  CEA, CA724 and CA199
Peripheral blood inflammatory index | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  The ratio of lymphocytes to monocytes (LMR) and ratio of Lymphocyte to neutrophil ratio (LNR)
Prognostic nutritional index | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  Serum albumin level (g/L) +5× total number of peripheral blood lymphocytes (×10 ^ 9 /L)
Quality of life of the patient | Before and after every cycle of treatment (each cycle is 28 days), assessed up to death or 3 years after surgery.
  This will be measured with Quality of Life Questionnaire of Stomach22 (QLQ-STO22). The minimum score is 22 and the maximum is 88. A higher score indicates a poorer quality of life.
Evaluation of the patient's symptoms | Before and after every cycle of treatment (each cycle is 28 days), assessed up to death or 3 years after surgery.
  This will be measured with M. D. Anderson Symptom Inventory (MDASI-GI) and Postgastrectomy Syndrome Assessment Scale (PGSAS-45). The minimum score of MDASI-GI is 0 and the maximum is 240. The minimum score of PGSAS-45 is 0 and the maximum is 271. A higher score indicates a poorer symptom.
Medication compliance | From randomization to the end of the sixth course of medication （up to 24 weeks）.
  The number of cases and percentage were calculated as < 80%, 80-120% and > 120%
Percentage of Participants With Adverse Events | Baseline until disease progression, death, or assessed up to 36 months after surgery.
  Percentage of Participants With Adverse Events in different arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Professor, Study Director — Guang 'anmen Hospital, China Academy of Chinese Medical Sciences; Yu Wu, Professor, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences; Shijie Zhu, Professor, Principal Investigator — Wangjing Hospital, China Academy of Chinese Medical Sciences; Hong Zhao, Professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Lizhu Lin, Professor, Principal Investigator — The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine; Ling Xu, Professor, Principal Investigator — Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine; Peng Shu, Professor, Principal Investigator — Jiangsu Hospital of Traditional Chinese Medicine
Locations (6):
- China (6):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Jiangsu Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be issued to publications through scientific journals and conference reports. The anonymized datasets used and/or analyzed during the current study are available from the sponsor-investigator on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Cao L, Zhu G, Wang X, Kuang Z, Song X, Ma X, Zhu X, Gao R, Li J. Yiqi Wenyang Jiedu prescription for preventing and treating postoperative recurrence and metastasis of gastric cancer: a randomized controlled trial protocol. Front Oncol. 2024 Jul 5;14:1326970. doi: 10.3389/fonc.2024.1326970. eCollection 2024. PMID 39035732